CLINICAL TRIAL: NCT00178802
Title: Phase II Study of Mild Whole Body Hyperthermia Combined With 5-Fluorouracil/Interferon-a/Liposomal Doxorubicin in Patients With Advanced Malignancy
Brief Title: Chemotherapy With Whole Body Hyperthermia to Treat Resistant Breast, Endometrial, Cervical and Ovarian Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Joan M.C Bull, M.D., The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-01-111; HSC-MS-01-111
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Breast Neoplasms; Endometrial Neoplasms; Cervix Neoplasms; Ovarian Neoplasms
Keywords: breast cancer; endometrial cancer; cervical cancer; ovarian cancer
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): thermochemotherapy using fever-range whole-body thermal therapy combined with continuous infusion 5-fluorouracil, Doxil, and low-dose interferon-alpha.
  Interventions: Other: thermochemotherapy (with 5-fluorouracil/interferon-a/liposomal doxorubicin)

INTERVENTIONS:
Other: thermochemotherapy (with 5-fluorouracil/interferon-a/liposomal doxorubicin) — 5-fluorouracil 400 mg/m2 i.v. over 24 hours for 5 days
  Doxil (liposomal doxorubicin) 40 mg/m2 over 1 hour
  Fever-range whole-body thermal therapy to 40 oC (104 oF) for 6 hours duration daily
  Low-dose interferon-alpha 100,000 i.u. s.c. daily for the duration of the protocol

SUMMARY:
Thermal therapy (hyperthermia of heat) can increase the effect of chemotherapy treatments. By itself, thermal therapy can also kill cancer cells. By using thermal therapy to treat the whole body, the investigators can treat cancer cells wherever they are throughout the entire body. In this study, the investigators are testing the combination of thermal therapy combined with chemotherapy to see:

1. if it improves the effect of the chemotherapy drugs,
2. if it helps the body fight the cancer cells, and
3. if this treatment is safe for the patient.

This study does not offer heat treatment alone. Any patient with advanced or metastatic breast, or endometrial cancer resistant to standard treatment may be treated with the phase II protocol therapy; however, the patient will need to undergo some medical tests to make sure this treatment would be safe for them.

DETAILED DESCRIPTION:
Once a patient has been accepted for this study, the patient will need to have a Central Venous line (CV line or port) if they do not already have one. (this may be placed by the patient's own doctor, or it can be done here).

The treatment cycle begins with a continuous 24-hour intravenous infusion of 5-Fluorouracil (5-FU) over a period of 5 days. This regimen will end 24 hours prior to the scheduled heat treatment. In addition, at the beginning of the treatment, the patient will begin daily, low-dose Interferon-alpha injections for the duration of their participation in this study. The drug, Interferon-alpha, is given to stimulate the immune system and to decrease tumor microvasculature. Interferon-alpha also interrupts the division of cancer cells and slows tumor growth.

The fever-range whole-body heat treatment is performed while the patient is under light conscious sedation. With this type of sedation, the patient is awake during the treatment but not uncomfortable. This type of sedation method is used to reduce the discomfort of the 6-hour heat treatment procedure yet allows the patient to respond to verbal commands.

The patient's body temperature is elevated to 40oC (104oF) over a period of 60-90 minutes. When the body reaches the target 40 oC, we will maintain that body temperature for six hours. At the conclusion of the six hours of heat treatment, the patient will be cooled to their normal body temperature, over 30-45 minutes. The Doxil chemotherapy will then be infused i.v. over a period of 2 hours.

The entire procedure lasts approximately 8-10 hours. After the treatment is completed, we observe the patient for 2 to 12 hours to make sure the treatment has been well tolerated.

The patient will continue the daily low-dose Interferon-alpha injections. Additionally, the patient will be given daily Leukine (sargramostim) cytokine injections usually beginning 3-5 days after receiving chemotherapy to help support the immune system by helping the body create more white blood cells, which are important in helping your body fight infection.

After treatment, the patient will need a complete blood count with platelet and differential count each week. These lab studies can be done at the patient's own doctor's office as long as the results are faxed to us. They can also be done in our clinic. The treatment cycle will be repeated every 28 days.

We always attempt to perform at least two thermochemotherapy cycles. After the second treatment, CT and/or MRI scans are repeated to see if the tumor has changed. These scans, along with a physical examination and the lab studies, are used to determine if additional heat treatments will be performed. Additional treatments continue based on how well a patient responds to the treatment. There is no limit to the number of heat treatments a patient may have.

ELIGIBILITY:
Inclusion Criteria:

* Resistant breast, endometrial, cervix, or ovarian cancer
* No active metastasis to the brain
* No more than 8 previous regimes of Doxil
* Successful completion of preliminary function tests
* Good ECOG score

Exclusion Criteria:

* Active metastasis to the brain
* 8 or more previous cycles of Doxil
* Poor completion of preliminary function tests
* Poor ECOG score

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1996-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 5 years
Response duration | 5 years

SECONDARY OUTCOMES:
Toxicity | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joan M Bull, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States